CLINICAL TRIAL: NCT05146804
Title: ''The PROtective Effect of SulforAphaNe on Chronic Low-grade Inflammation in Healthy Participants'': The PRO SANI Study
Brief Title: The PROtective Effect of SulforAphaNe on Chronic Low-grade Inflammation in Healthy Participants
Acronym: PRO SANI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Prevention
Other Study IDs: PRO SANI NL77272.068.21
Record Dates: First submitted 2021-11-15; First posted 2021-12-07 (Actual); Last update posted 2022-04-13 (Actual); Status verified 2022-04

CONDITIONS: Inflammation
Keywords: Sulforaphane Inflammation Challenge BroccoCress; Inflammation; Challenge; BroccoCress
MeSH Terms: conditions — Inflammation | interventions — sulforaphane

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BroccoCress/Affilla Cress (Other): Potential participants will be screened after showing their interest to participate to the study. When they are considered eligible to participate (after a phone call with the executing researcher), participants will be randomized into one of the two groups in this study: either consuming the broccoli sprouts on day one (visit 1) and the placebo product in the second visit, or the other way around (placebo product on day 1 and the intervention during the second visit). Both days, participants will consume the PhenFlex, the challenge product with the high caloric load. This will allow for analyzing the effectiveness of the intervention on different biomarkers of chronic, low-grade inflammation, with the main objective being on endothelial activation.
  Interventions: Other: BroccoCress; Other: Affilla Cress
- Affilla Cress/Broccocress (Other): Potential participants will be screened after showing their interest to participate to the study. When they are considered eligible to participate (after a phone call with the executing researcher), participants will be randomized into one of the two groups in this study: either consuming the broccoli sprouts on day one (visit 1) and the placebo product in the second visit, or the other way around (placebo product on day 1 and the intervention during the second visit). Both days, participants will consume the PhenFlex, the challenge product with the high caloric load. This will allow for analyzing the effectiveness of the intervention on different biomarkers of chronic, low-grade inflammation, with the main objective being on endothelial activation.
  Interventions: Other: BroccoCress; Other: Affilla Cress

INTERVENTIONS:
Other: BroccoCress — BroccoCress® is a brand name for an edible plant, broccoli sprouts. BroccoCress® is a product within the group of vegetable sprouts.
  Other Names: Sulforaphane
Other: Affilla Cress — Pea sprouts commercially available as Affilla Cress® will be used as placebo in this study since these sprouts do not contain Glucoraphanin/Sulforaphane.
  Other Names: Pea sprouts

SUMMARY:
Rationale:

Most non-communicable diseases are partially affected by low-grade chronic inflammation. Research has shown that sulforaphane, an ingredient found in abundance in broccoli, shows promise as a potent anti-inflammatory substance. However, its potential in the settings of the caloric-induced inflammatory response has not been tested.

Objective:

In the present study, the investigators aim to assess the efficacy of sulforaphane on biomarkers of inflammation and other markers of phenotypic flexibility in healthy participants subjected to the standardized 'PhenFlex' challenge. Study design: Double-blind, crossover, randomized, placebo-controlled, intervention study.

Study population: Healthy human volunteers (18-50 years old) Intervention: Participants will receive 16 grams (intervention) of broccoli sprouts (BroccoCress®) and 16 grams of Affilla Cress® (placebo) on different occasions in randomized order.

Main study parameters/endpoints: The main endpoint of the present study is to demonstrate that sulforaphane can influence endothelial activation measured as changes in plasma concentrations of sVCAM and sICAM in a caloric challenge test in healthy participants. Nature and extent of the burden and risks associated with participation, benefit and group relatedness: Use of BroccoCress® in human subjects has not been related to adverse effects, except of the individuals who show individual intolerance to cruciferous vegetables. Those individuals will not be permitted into the study. The 'PhenFlex', a high-fat, high-glucose, high-calorie drink, is used for the caloric load. The PhenFlex has been used in three studies before, with no side effects reported after consumption. Sampling of venous blood can potentially cause complications (haematoma formation, fainting, etc). The procedures involved in this study will include an interview, assessment of vital signs, completion of the study related questionnaires and collection of blood and urine samples. Volunteers will receive an unsubstantial financial reward for the participation in this study. The results will provide information on whether the intake of cruciferous vegetables rich in sulforaphane can increase resilience to excessive inflammatory stimuli associated with caloric overload and potentially provide evidence on the role of dietary ingredients in combating chronic low-grade inflammation.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent form (ICF) prior to initiation of any study related procedures
* Male or female volunteer
* Age 18-50 years
* BMI between 18.5-30 kg/m2
* Stable weight and no intention to lose weight until completion of the study; no reported weight loss or weight gain of ≥ 5 kg 3 months prior to inclusion into this study
* Constant eating habits during at least 3 months prior to inclusion into the study

Exclusion Criteria:

* Having a history of medical or surgical events that may significantly affect the study outcomes and inflammatory response. More specifically, the previous diagnosis of an inflammatory condition or disease or a history of hypothyroidism, chronic kidney or/and liver disorders, coronary artery disease, malignant hypertension, seizures.
* Involved in intensive sports activities more than 4 times a week or at top sport level (e.g. playing football, tennis, running, race-cycling, swimming)
* Regular intake of medication. More specific, medication that may affect inflammatory response including NSAIDs such as Ibuprofen, Naproxen, Diclofenac is not allowed from 2 weeks before screening until the end of the study. Participants are allowed to use oral contraceptives before and during the study.
* Psychotic, addictive or other mental disorders limiting the ability to provide informed consent or to comply with the study requirements
* Aversion, intolerance or allergy to cruciferous vegetables (e.g. kale consumption; bloating) or ingredients of the PhenFlex drink (palm olein, dextrose, protein supplement, vanilla aroma).
* Use of dietary supplements with potential effects on antioxidant or inflammatory status within 4 weeks prior to inclusion into this study. Examples of dietary supplements not allowed in the study include supplements containing flavonoids, glucosinolates, carotenoids, ergothioneine, polyacetylenes and polysaccharides. - Excessive alcohol consumption (≥ 28 consumptions approx. 250 g alcohol per week)
* Viral or bacterial infection requiring use of antibiotics, laxatives and anti-diarrheal drugs within 4 weeks prior to inclusion into this study
* Pregnancy and/or breastfeeding
* Reported slimming or medically prescribed diet
* Vegetarian or vegan lifestyle

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2021-11-11 (Actual); Primary Completion 2022-02-03 (Actual); Study Completion 2022-02-03 (Actual)

PRIMARY OUTCOMES:
Change of endothelial activation. | Day 1, Day 8±3
  Change of plasma concentrations of sVCAM (ng/mL) and sICAM (ng/mL)

SECONDARY OUTCOMES:
Change of the systemic low-grade inflammation score (SIS) | Day 1, Day 8±3
  The systemic low-grade inflammation score (SIS). The SIS score will be constructed from:
  * Biomarkers that represent metabolic tissue inflammation (IL-1b,IL-6,and tumor necrosis factor alpha [TNF-a])
  * Biomarkers of immune cell recruitment (C-C motif ligand-2[CCL-2]),IL-8, soluble intercellular adhesion molecule-1 [sICAM-1], soluble vascular cell adhesion molecule-1 [sVCAM-1])
  * Biomarkers of inflammation resolution(IL-10, adiponectin)
  * Biomarkers of overall inflammation (CRPandIL-12p70).
  A SIS will be generated summing the z-score log-transformed inflammatory biomarkers plasma concentration (CRP, IL-1 b, IL-6, IL-8, IL-12 p70, TNF-a, CCL-2, sICAM-1, and sVCAM-1). The Z-score log-transformed plasma adiponectin and IL-10 levels will be subtracted from SIS because of their well-known anti-inflammatory functions.
Change of NF-κB activity and Nrf2 activity. | Day 1, Day 8±3
  NF-KB activity and Nrf2 activity will be measured by ELISA to assess pathway activation.
  Detection principle of Human Nuclear Factor Kappa B ( NF-κB)ELISA kit This experiment use double-sandwich elisa technique and the ELISA Kit provided is typical.
  The Human NRF2 ELISA Kit is a solid-phase sandwich Enzyme-Linked Immunosorbent Assay (ELISA) designed to detect and quantify the level of human NRF2 in cell culture supernatants, plasma, and serum.
Change of urinary concentrations (μmol) of SFN and metabolites will be determined; SFN-glutathione, SFN-cysteine-glycine, SFN-cysteine, and SFN-N-acetylcysteine (SFN-NAC). | Day 1, Day 8±3
  Estimation of bioavailability
Change of Urinary 11dhTxB2. | Day 1, Day 8±3
  Quantification of urinary 11dhTxB2 (μg) by ELISA
Change of HRV | Day 1, Day 8±3
  HRV will be assessed in short term (5 min) ECG recording obtained in supine position and analysed as recommended by current standards (ESC / NASPE, 1996). Total power (TP), high-frequency power (HF), low frequency power (LF), and very low- frequency power (VLF) will be derived from the spectral analysis. Also, the following time domain indices will be assessed: standard deviation of normal RR intervals (SDNN); square root of the mean squared differences of successive RR interval, (RMSSD); percentage of differences between adjacent normal RR intervals exceeding 50 milliseconds (pNN50). The recordings of ECG will be performed 4 times: (i) before administration of investigational product; (ii) before administration of PhenFlex; (iii) 30 min after administration of PhenFlex; (iv) 2 hours administration of PhenFlex.

CONTACTS AND LOCATIONS:
Locations (1):
- Campus Venlo, Maastricht University, Venlo, Limburg, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] van Steenwijk HP, Vinken A, van Osch FHM, Peppelenbos H, Troost FJ, Bast A, Semen KO, de Boer A. Sulforaphane as a potential modifier of calorie-induced inflammation: a double-blind, placebo-controlled, crossover trial. Front Nutr. 2023 Nov 28;10:1245355. doi: 10.3389/fnut.2023.1245355. eCollection 2023. PMID 38089924
- [Derived] van Steenwijk HP, Winter E, Knaven E, Brouwers JF, van Baardwijk M, van Dalum JB, Luijendijk TJC, van Osch FHM, Troost FJ, Bast A, Semen KO, de Boer A. The beneficial effect of sulforaphane on platelet responsiveness during caloric load: a single-intake, double-blind, placebo-controlled, crossover trial in healthy participants. Front Nutr. 2023 Jul 6;10:1204561. doi: 10.3389/fnut.2023.1204561. eCollection 2023. PMID 37485383